CLINICAL TRIAL: NCT01915121
Title: An Educational Intervention for Patients With Bladder Cancer 121193-MRSG-11-103-01-CPPB American Cancer Society
Brief Title: An Educational Intervention for Patients With Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 09-0479
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Intervention; Education; Randomized Controlled Trials
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Early Intervention, Educational; Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Intervention (Active Comparator): In this session, participant will be provided with information about bladder cancer treatment options, and training tools directly related to Bladder Cancer.
  Interventions: Behavioral: Education Intervention
- Nutrition Intervention (Placebo Comparator): In this session, participant will be provided with information about nutrition information directly related to bladder cancer recovery
  Interventions: Behavioral: Nutrition Intervention

INTERVENTIONS:
Behavioral: Education Intervention — 1-hour educational and training sessions. In this session, participant will be provided with information about bladder cancer treatment options, and training tools directly related to Bladder Cancer. In 4 to 5 days following the session, participants will be asked to schedule the time to talk about experience and how the intervention affects their treatment decision making and to answer some questions about the educational and training session they attended. Participants will then be called after 1-month, 3-month, and 6-month after their bladder cancer treatment to follow up.
  Arms: Education Intervention
Behavioral: Nutrition Intervention — 1-hour educational and training sessions. In this session, participant will be provided with nutrition information directly related to Bladder Cancer recovery. In 4 to 5 days following the session, participants will be asked to schedule the time to talk about experience and how the intervention affects their treatment decision making and to answer some questions about the educational and training session they attended. Participants will then be called after 1-month, 3-month, and 6-month after their bladder cancer treatment to follow up.
  Arms: Nutrition Intervention

SUMMARY:
The study main objectives are to enhance treatment decision making and improve quality of life and post-treatment health care among patients diagnosed with invasive bladder cancer.

Bladder cancer (BL Ca) is the 5th most commonly diagnosed cancer in the US . BL Ca is more common among men than women and 90% of all patients are over the age of 55. Surgery to remove the bladder followed by one of three diversion techniques (i.e., ileal conduit, continent reservoir, and neobladder) is the standard therapy following invasive bladder cancer. The emotional, functional, physical, and social impact of invasive Bl Ca treatment on patients' QOL and adjustment can be devastating. This impact significantly varies by treatment option. Treatment decision making in for BL Ca is difficult at best and potentially susceptible to a number of cognitive and affective factors (e.g., patients' emotional reaction, values, and expectations). Thus, in addition to adjusting to a potential life-threatening disease, having to cope with uncertainty about the efficacy and outcomes of different treatment options adds to the overall distress and may impair effective decision-making. In spite of increasing efforts in health communication and patient education, no study has examined treatment decision making among invasive bladder patients or has provided an educational intervention to facilitate treatment decision making among this population. To this end, and guided by the Self-Regulation theory (SRT) that emphasizes the role of cognitive and emotional factors in decision making, we have designed and pilot tested the acceptability of a preliminary educational and training experiential intervention (ETE) to address this gap in the literature. The ETE intervention uses new and innovative educational strategies and methods to educate patients about their treatment options and to facilitate their treatment decision making.

DETAILED DESCRIPTION:
The goals of the study are: 1) to further enhance the design and application of the ETE intervention, and 2) to provide data on the efficacy of the refined ETE intervention in a randomized-controlled study (RCT). To achieve these 2 goals, the study is divided in to 2 phases.

PHASE 1: To enhance and refine the design and application of the preliminary ETE intervention:

Aim 1-a: To explore knowledge, beliefs, values and expectations about treatment options, treatment decision making, and quality of life (QOL) among patients with BL Ca.

To achieve Aim 1-a of Phase 1, as a first step, 2 focus groups (FG; N = 10 each) of invasive BL Ca patients will be conducted to a) examine knowledge, beliefs, values, expectations, and affective responses about treatment options and treatment decision making, b) record difficulties and problems in post-surgical health care (e.g., using stoma appliances and catheters), and c) explore concerns patients have as they live with the impact of treatment. The ETE intervention will be refined based on FG results.

Aim 1-b: To explore patients' acceptability of the refined ETE intervention. To achieve Aim 1-b of Phase 1, additional 2 FG (FG; N = 10 each) of BL Ca survivors will be conducted to solicit input about the design and acceptability of the refined ETE intervention.

PHASE 2: Aim 2. To assess the efficacy of the ETE intervention in small RCT To achieve Aim 2 of Phase 2, a two-group RCT (standard care (SC) plus time and attention control condition, N = 62 patients; SC plus ETE intervention N = 62 patients) will be conducted to examine the efficacy of the ETE intervention. Phase 2 will provide a) a test of the efficacy of the refined ETE intervention for reducing decisional conflict and regret, and improving QOL and post-treatment stoma and pouch care controlling for potential clinical and socio-demographic covariates (e.g., treatment type, age).

ELIGIBILITY:
Phase 1 (Focus groups/ In-depth Interview)

Inclusion Criteria:

* treatment of invasive Bladder Cancer a with cystectomy and one of the three major urinary diversion methods
* English speaking
* between the ages of 18 and 85
* able and willing to provide informed consent
* may have received neoadjuvant or adjuvant chemotherapy, radiation therapy, and immunotherapy (BCG)

Exclusion Criteria:

* metastatic disease or cancer recurrence
* presence of other primary cancers
* no access to a telephone

Phase 2 (randomized-controlled-study)

Additional Exclusion Criteria:

- treatment decision is made and /beginning/completion of treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Decisional Regret Scale | Baseline
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 1 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 3 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 6 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Self-Efficacy Scale | Baseline
  The intervention is designed to enhance treatment decision making.
Decisional Self-Efficacy Scale | 1 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Self-Efficacy Scale | 3 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Self-Efficacy Scale | 6 month follow up
  The intervention is designed to enhance treatment decision making.
Treatment-related Values | Baseline
  The intervention is designed to enhance treatment decision making.
Treatment-related Values | 1 month follow up
  The intervention is designed to enhance treatment decision making.
Treatment-related Values | 3 month follow up
  The intervention is designed to enhance treatment decision making.
Treatment-related Values | 6 month follow up
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | Baseline
  Bladder Cancer knowledge Scale
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 1 month follow up
  Bladder Cancer knowledge Scale
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 3 month follow up
  Bladder Cancer knowledge Scale
  The intervention is designed to enhance treatment decision making.
Decisional Regret Scale | 6 month follow up
  Bladder Cancer knowledge Scale
  The intervention is designed to enhance treatment decision making.

SECONDARY OUTCOMES:
quality of life | Baseline
  FACT-BL, Emotional, physical, function, and social Wellbeing Subscales
quality of life | 1 month follow up
  FACT-BL, Emotional, physical, function, and social Wellbeing Subscales
quality of life | 3 month follow up
  FACT-BL, Emotional, physical, function, and social Wellbeing Subscales
quality of life | 6 month follow up
  FACT-BL, Emotional, physical, function, and social Wellbeing Subscales
post-surgical self-care | Baseline
  FACT-BL Ca additional concern
post-surgical self-care | 1 month follow up
  FACT-BL Ca additional concern
post-surgical self-care | 3 month follow up
  FACT-BL Ca additional concern
post-surgical self-care | 6 month follow up
  FACT-BL Ca additional concern
CES-D scale Illness Perception Questionnaire (IPQ) | Baseline
CES-D scale Illness Perception Questionnaire (IPQ) | 1 month follow up
CES-D scale Illness Perception Questionnaire (IPQ) | 3 month follow up
CES-D scale Illness Perception Questionnaire (IPQ) | 6 month follow up
Cancer worries scale | Baseline
Cancer worries scale | 1 month follow up
Cancer worries scale | 3 month follow up
Cancer worries scale | 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nihal E Mohamed, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - James J. Peters VA Medical Center, The Bronx, New York